CLINICAL TRIAL: NCT03437421
Title: Effect of Vitamin D Supplementation on Myocardial Regional Function by Dobutamine Stress Echocardiography in Diabetic Patients.
Brief Title: Myocardial Function and Vitamin D Supplementation in Diabetes.
Acronym: VitaDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UAPV-022018-SFC
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Complications; Vitamin D Deficiency; Vitamin D Supplementation; Myocardial Dysfunction
Keywords: myocardial function; vitamin D; stress echocardiography; diabetes
MeSH Terms: conditions — Diabetes Complications; Vitamin D Deficiency; Diabetes Mellitus | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Type I and II diabetic patients will be investigated. Within each diabetic population, vitamin D deficient and non-deficient individuals will be compared at baseline. Then, within each diabetic population, those with vitamin D deficiency at baseline will be compared before and after a 3 month vitamin D supplementation.
Who Masked: Outcomes Assessor
Masking Description: Single-masked study. Clinicians and researchers in charge of main outcomes (eg cardiac remodelling and global function, regional myocardial function) measurements will not be aware of group allocation (eg vitamin D deficient and non-deficient sub-groups) and time study (eg baseline or post vitamin D supplementation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type II diabetic patients (Experimental): 3 month Vitamin D3 (cholecalciferol) supplementation in patients with vitamin D deficiency, based on 25-OH-D3 dosage.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Type I diabetic patients (Experimental): 3 month Vitamin D3 (cholecalciferol) supplementation in patients with vitamin D deficiency, based on 25-OH-D3 dosage.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — * Patients with 29≤ 25-OH-D3 ≥20 ng/mL will receive 200 000 UI orally the first month (100 000 UI at T0 + 100 000 UI at T0+15 days, UVEDOSE™ Laboratoires Crinex, Montrouge, France) followed for the last 2 months by one daily dose (5 drops orally = 1 000 UI/day, DÉDROGYL™ , DB Pharma, La Varenne-Saint-Hilaire, France).
  * Patients with : 19≤ 25-OH-D3 ≥10 ng/mL will receive orally 300 000 UI (100 000 UI at T0 + 100 000 UI at T0+23days + 100 000 UI at T0+45days; UVEDOSE™) followed for the last month by one daily dose (5 drops orally =1 000 UI/day, DÉDROGYL™ ).
  * Patients with : 25-OH-D3 <10 ng/mL will receive orally 400 000 UI (100 000 UI at T0 + 100 000 UI at T0+15days + 100 000 UI at T0+30 days + 100 000 UI at T0+45days, UVEDOSE™) followed for the last month by one daily dose (5 drops orally =1 000 UI/day, DÉDROGYL™).

SUMMARY:
Vitamin D deficiency is recognized as a cardiovascular risk factor. Diabetic patients are of major risk for cardiovascular diseases and typically present with Vitamin D deficiencies. Myocardial function is altered in both type I and II diabetic patients but no data is today available on the effect of Vitamin D supplementation.

The aim of the study will be to investigate myocardial function (by deformation imaging techniques) at rest and during low-dose dobutamine stress echocardiography in both type I and II diabetic patients. Within each diabetic population, myocardial function will be compared at baseline between the vitamin D deficient and non-deficient individuals. Furthermore, the investigators will study the effect of a 3 month supplementation in those with deficiencies.

DETAILED DESCRIPTION:
Rationale:

Vitamin D exerts a principal role in homeostasis of calcium and phosphorus. However, recent studies indicated also its important function in cell differentiation, proliferation and growth as well as regulation of the immune system.

Vitamin Deficiency is today recognized as a risk factor for cardiovascular disease (CVD). Diabetic patients are of major risk for CVD. They typically present with Vitamin D deficiencies. Experimental studies have established as a result of Vitamin D deficiency alterations in intrinsic cardiac contractile and relaxation properties, hypertrophy and fibrosis. Regional myocardial function is altered in both type I and II diabetic patients. In type II diabetic individuals, myocardial dysfunction is furthermore exacerbated in those with Vitamin D deficiency compared to those with normal levels. In patients free from CV risk and deficient in Vitamin D, regional myocardial function improved after Vitamin D supplementation. To the best of our knowledge, no scientific study is today available on the effect of Vitamin D supplementation on regional myocardial function in diabetic patients deficient in vitamin D.

Objectives and Methodology:

* To compare regional myocardial linear deformation and torsion, at rest and in response to a DB stress in diabetic patients deficient and non-deficient in Vitamin D.
* To evaluate the impact of vitamin D supplementation in those with vitamin D deficiency.

All the diabetic patients will benefit from a clinical (medical history, drug therapy, ECG, blood pressure, ...), anthropometric (abdominal obesity indices) and biological (carbohydrate and lipid balance, markers of inflammation and heart failure, vitamin D glucose and insulin status) evaluation. In addition, conventional echocardiography (remodelling and global diastolic and systolic function) complemented by a functional analysis by tissue Doppler imaging will be performed. Furthermore, 2D cine loops will be recorded in the apical 4, 3 and 2- chamber views for the assessment of regional myocardial longitudinal deformations as well as in the parasternal short axis (base, mid and apex) for the evaluation of circumferential deformations and basal and apical rotation and torsion, at rest and under low dose dobutamine (110 and 120 bpm).

Vitamin D supplementation:

Patients with vitamin D deficiency will be investigated before and after a 3 month cholecalciferol supplementation.

For this purpose 25-OH-D3 with be evaluated at baseline.

* Patients with 29≤ 25-OH-D3 ≥20 ng/mL will receive 200 000 UI orally the first month (100 000 UI at T0 + 100 000 UI at T0+15 days, UVEDOSE™ Laboratoires Crinex, Montrouge, France) followed thereafter for the last 2 months by one daily dose (5 drops orally = 1 000 UI/day, DÉDROGYL™ , DB Pharma, La Varenne-Saint-Hilaire, France).
* Patients with : 19≤ 25-OH-D3 ≥10 ng/mL will receive orally 300 000 UI (100 000 UI at T0 + 100 000 UI at T0+23days + 100 000 UI at T0+45days; UVEDOSE™ Laboratoires Crinex, Montrouge, France) followed thereafter for the last month by one daily dose (5 drops orally =1 000 UI/day, DÉDROGYL™ , DB Pharma, La Varenne-Saint-Hilaire, France).
* Patients with : 25-OH-D3 <10 ng/mL will receive orally 400 000 UI (100 000 UI at T0 + 100 000 UI at T0+15days + 100 000 UI at T0+30 days + 100 000 UI at T0+45days, UVEDOSE™ Laboratoires Crinex, Montrouge, France) followed thereafter for the last month by one daily dose (5 drops orally =1 000 UI/day, DÉDROGYL™ , DB Pharma, La Varenne-Saint-Hilaire, France).

ELIGIBILITY:
Inclusion Criteria:

• Male and female 40-65 years old, asymptomatic and free from epicardial coronary artery disease.

Exclusion Criteria:

* body mass index > 35 kg / m2, defining severe obesity,
* Under insulin therapy (for Type II only)
* Poorly controlled hypertension (> 140/95)
* LV ejection fraction (LVEF) < 55%
* Peripheral vascular disease (> stage II of Leriche)
* Heart disease or known coronary artery disease,
* Known and poorly compensated thyroid dysfunction,
* Nocturnal apnea syndrome,
* Inability to give written informed consent,
* Chronic diseases,
* moderate to severe left ventricular hypertrophy :> 109 g / m2 in women and> 132 g / m2 in men and parietal thickness > 13mm.
* poor glycemic control (HbA1c > 9%)
* poor echogenicity
* severe autonomic or peripheral neuropathy,
* Severe diabetic retinopathy,
* Advanced Diabetic nephropathy (defined by documented proteinuria and/or renal failure).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-19 (Actual)

PRIMARY OUTCOMES:
Change in longitudinal strain | Before and after 3 month of Vitamin D supplementation
  Index of myocardial function measured using deformation imaging technique by echocardiography, at rest and under dobutamine stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Henri Duffaut, Avignon, PACA, France

REFERENCES:
- [Derived] Obert P, Nottin S, Philouze C, Aboukhoudir F. Major impact of vitamin D3 deficiency and supplementation on left ventricular torsional mechanics during dobutamine stress in uncomplicated type 2 diabetes. Nutr Metab Cardiovasc Dis. 2023 Nov;33(11):2269-2279. doi: 10.1016/j.numecd.2023.06.017. Epub 2023 Jun 24. PMID 37543521